CLINICAL TRIAL: NCT03513783
Title: Elbow Extension Restoration Surgery in People With Tetraplegia: Evolution of the Muscular Co-activations of the Upper Limb During the Post-operative Rehabilitation MouvSupReaTetra
Brief Title: Elbow Extension Restoration Surgery in People With Tetraplegia: Evolution of the Muscular Co-activations of the Upper Limb During the Post-operative Rehabilitation
Acronym: MouvSupReaTetr
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: not enough patients
Sponsor: Nantes University Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: RC17_0466
Record Dates: First submitted 2018-04-10; First posted 2018-05-02 (Actual); Last update posted 2023-12-14 (Actual); Status verified 2023-12

CONDITIONS: Tetraplegia
Keywords: Spinal Cord Injury; tendon transfer; muscle synergy; muscle co-activation; electromyography
MeSH Terms: conditions — Quadriplegia; Spinal Cord Injuries

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: measurement of human movement — The objective measurement of human movement through the use of kinematic markers and electromyography is a clinical exam commonly performed to analyze the movements of patients with motor control disorders. The different steps are the following:
  * A clinical exam is performed by the Physical Medicine & Rehabilitation clinician (passive range of motion , spasticity, muscular force, etc.).
  * Intramuscular and surface electromyography and kinematic markers are placed on the upper limb of the participant. A maximum of two intramuscular electrodes will be inserted with guiding of an echography system.
  * The participant will be asked to perform several upper limb movements: specifically, he will be asked to perform consecutive cycles of elbow extension-flexions with the shoulder at different levels of abduction. Times of rest will be given to the participants.
  Time of the procedure is estimated to 1h, with only about 2 minutes of active effortless movements from the participants.

SUMMARY:
Patients with C5 or C6 tetraplegia have paralysis of the triceps brachii. Elbow extension can be surgically restored by transferring the tendon from a preserved muscle onto the tendon of the paralyzed triceps brachii.

The most frequently used method transfers the posterior deltoid tendon. However, transferring the posterior deltoid can create an imbalance in the shoulder joint and this technique is not recommended when the clavicular head of the pectoralis major is weak.

In such cases, a preferred method is a biceps brachii tendon transfer. The success of this intervention relies on the ability of the patient to dissociate the drive between the transferred biceps brachii and the other elbow flexor muscles.

Even though tendon transfers are widely used, the subsequent reorganization of muscle coordination strategies remains largely unknown. The identification of muscle synergies and co-coactivations from electromyography (EMG) signals, defined as groups of muscles activated in synchrony, may help to provide a deeper understanding of changes in muscle coordination. The objective of this study is to investigate for the first time the reorganization of muscle coordination after surgical restoration of elbow extension through the identification of muscle synergies and the quantification of muscle co-activations.

Four participants with tetraplegia will take part to this study. The experimental procedure will be conducted before their surgery and once a month during 6 months after their surgery.

The procedure consists of performing consecutive elbow extension-flexion cycles with the shoulder abducted at different angles. Surface and intramuscular EMG measurements will be collected for several upper limb muscles. Muscle synergies and co-activations will be extracted from the EMG measurements.

DETAILED DESCRIPTION:
There is a need for a detailed and quantified follow-up during rehabilitation after an elbow extension restoration in people with tetraplegia. Surface or intramuscular electromyography (EMG) gives information on muscular activation, and can detect small but clinically relevant modifications in muscular activation of patients with tetraplegia. To this day, no study measured the evolution of muscular activation in the upper limb of people with tetraplegia who underwent an elbow extension restoration surgery. The objective of this study is to investigate for the first time the reorganization of muscle coordination after surgical restoration of elbow extension through the identification of muscle synergies and the quantification of muscle co-activations.

Four participants with tetraplegia will take part to this study. The experimental procedure will be conducted before their surgery and once a month during 6 months after their surgery.

The 1h procedure consists of performing consecutive elbow extension-flexion cycles with the shoulder abducted at different angles. Surface and intramuscular EMG measurements will be collected for several upper limb muscles. Kinematic markers will be placed in order to measure the upper limb range of motion and movement velocity.

Surface EMG signals will be band-pass filtered (10-450Hz), full wave rectified, and smoothed with a low-pass filter (10Hz). Onset and offset times will be defined through the calculation of an activation threshold. For each session and each muscle, EMG amplitude will be normalized to its peak value across all trials. Each elbow extension-flexion cycle will be interpolated to 100 time points: 0-50% was extension; 50-100% flexion.

For each participant and each movement, all combinations of muscle synergies will be identified using non-negative matrix factorization (NMF) from the EMG data and data will then be averaged across the cycles. Co-activations will be directly identified from the EMG data.

ELIGIBILITY:
Inclusion Criteria:

* Participants are min 18 years old.
* Participants have a tetraplegia level C5 or C6
* Participants are hospitalized at Saint Jacques hospital
* Participants are candidates to an elbow extension restoration surgery.
* Participants have health insurance

Exclusion Criteria:

* Participants are unable to understand or follow instructions.
* Participants are under guardianship
* Participants are under anti-thrombotic therapy
* Participants are pregnant

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 3 (Actual)
Dates: Start 2018-09-10 (Actual); Primary Completion 2021-05-12 (Actual); Study Completion 2023-09-10 (Actual)

PRIMARY OUTCOMES:
Evolution of muscular co-activations with time | Before and one a month for 6 months after the surgery.
  The primary outcome measure of interest is the evolution of the muscular co-activations after the restoration surgery. Muscular co-activations represent the simultaneous activation of two or more muscles (unit %). It will be plotted against time (unit in months).

SECONDARY OUTCOMES:
Evolution of the extension range of motion | Before and one a month for 6 months after the surgery.
  The secondary outcome measure of interest is the evolution of the range of motion after the restoration surgery. The range of motion (unit °) is extracted from the kinematic data obtained through the use of markers and motion capture. It will be plotted against time (unit in months).

CONTACTS AND LOCATIONS:
Locations (1):
- CHU de Nantes, Nantes, France